CLINICAL TRIAL: NCT04054141
Title: TMS for Treatment of Spasticity in Patients With MND
Brief Title: rTMS in Treatment of Spasticity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not meet target enrollment
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0434
Record Dates: First submitted 2018-08-13; First posted 2019-08-13 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: ALS

STUDY DESIGN:
Intervention Model Description: Open label rTMS treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- rTMS arm (Experimental): Each patient's participation will last a maximum of 12 weeks and involves 2 sessions of neurophysiological testing (TMS) sessions and 15 neurophysiological treatment sessions (rTMS).
  Patients will have a neurophysiological testing session (TMS) at the screening visit (week 0). Patients will then return for 15 neurophysiological treatment sessions (rTMS) within 14 days of screening. Patients must complete three neurophysiological treatment sessions (rTMS) during weeks 1, 2, 3, 4 and 5. The second neurophysiological testing session will be done at the final visit (week 5). Follow-up visits will be scheduled at weeks 7 and 10 (+/- 3 days). That is, the follow-up visits will occur two and five weeks after the final rTMS session which occurs on day 15.
  Interventions: Device: Mag Stim

INTERVENTIONS:
Device: Mag Stim — rTMS

SUMMARY:
This is an open-label clinical trial to determine the safety and efficacy of rTMS in reducing spasticity and improving quality of life among patients with upper motor neuron predominant motor neuron disease (MND).

DETAILED DESCRIPTION:
The study's objective is to evaluate the role of rTMS for symptom reduction of spasticity among patients with upper motor neuron predominant motor neuron disease. This study is 12-week open label safety and efficacy trial. A total of 10 subjects with PLS and UMN/ MND will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18, men or woman
* Diagnosis of upper motor neuron predominant ALS, which also includes patients with primary lateral sclerosis (PLS), as defined as only upper motor neuron features in at least 2 body segments.
* EMG within 3 months of enrollment with minimal or no evidence of lower motor neuron disease.
* Time from symptom onset > 18 months
* On a stable dose of, or has not taken, Riluzole for at least thirty days.
* Has not taken, or has received at least 2 cycles of dosing of, Edaravone prior to screening.
* Able to communicate clearly the desire to withdraw from the procedure at any stage.
* Impaired walking as measured by a Hauser Ambulation index of greater than 1 and less than 7 (2 to 6, inclusive).
* MMSE ≥ 22 and deemed by the PI as being capable of providing informed consent and following trial procedure.
* Has spasticity, equal or above 1 in the Ashworth Scale for spasticity in 2 or more muscle group of at least 3 months duration.
* Absence of exclusion criteria.

Exclusion criteria

* Patient has a history of drug or alcohol abuse within the past year;
* Patient has clinically significant abnormal laboratory values.
* Any concomitant disease or disorder that has spasticity-like symptoms or that may influence the subject's level of spasticity
* Received Botulinum Toxin during the preceding 6 months
* Bedridden and patients with tracheostomy.
* Fixed-tendon contractures
* Poorly controlled epilepsy or recurrent seizures (Subjects who have had one or more seizures in the year prior to Visit 1 will be excluded)
* Unable to provide an informed consent
* Unable to comply with the procedures
* Unable to communicate clearly if the subject wants to withdraw from the procedure at any stage
* History of brain surgery for any indication
* Has pacemaker, cochlear implants, brain stimulators, infusion pumps, intracardiac lines, metallic clips, other implanted electronic or ferroelectric metallic devices above the neck (Dental implants are permitted), piercing or body modification above the neck, known history of TMS related complications or side effects.
* MMSE <22.
* Female patients of child bearing period who are not practicing contraception.
* Female patients who are pregnant.
* Inability to perform either rTMS due to insufficient MEP amplitude (< 50 µv).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
safety of rTMS in subjects with PLS/UMN/MND. Number of participants with treatment related AE's will be measured with stringent stopping rules and reported. We hypothesize that no serious treatment related adverse event. | from week 0 to the end of the study, an average of 5 months.
  Transcranial magnetic stimulation is a non-invasive procedure used to stimulate small regions of the brain. The effect of rTMS on spasticity was studied in patients with stroke, MS, SCI and CP and found to be safe (4). There are no studies assessing safety of rTMS in patients with PLS and UMN/ MND with spasticity. Because it is so well tolerated in other diseases, we anticipate no adverse effects. However, we will systematically assess all adverse effects with stringent stopping rules for individual patients and the study. We hypothesize that no patient will have a serious treatment related adverse event. Therefore we will track the number of Participants With Treatment-Related AE as Assessed by CTCAE v4.0

SECONDARY OUTCOMES:
To evaluate efficacy of rTMS using a modified FDA approved protocol in research subjects with PLS and UMN/MND. | From week 0 to end of the study, an average of 5 months
  The secondary objective of this study is to determine if rTMS causes an improvement in walking speed in patients with PLS and UMN/MND. This will be determined by evaluation of subject's walking speed during treatment and for period after the rTMS stimulation series has stopped. The primary end point will be measured through the consistent improvement in the Timed 25 Foot walk test (T25FW).

CONTACTS AND LOCATIONS:
Locations (1):
- Shara Holzberg, New York, New York, United States